CLINICAL TRIAL: NCT00621946
Title: Escitalopram in the Treatment of Outpatients With Severe Asthma and Moderate or Severe Major Depressive Disorder: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Treatment of Outpatients With Severe Asthma and Moderate or Severe Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Sherwood Brown, Principal Investigator, MD/PhD, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 092007-057
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Results first posted 2013-12-27 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Severe Asthma; Moderate or Severe Major Depressive Disorder
Keywords: Asthma; Depression; Escitalopram
MeSH Terms: conditions — Asthma; Lymphoma, Follicular; Depressive Disorder, Major; Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Placebo Matching Escitalopram given orally daily (for a 12-week duration).
  Interventions: Drug: Placebo
- Escitalopram (Active Comparator): Once daily oral administration (for a 12-week duration) of 10 mg escitalopram tablets with an increase to 20 mg in those with a less than 30% decrease in HAM-D scores at week 4.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Placebo — Placebo Matching Escitalopram
  Other Names: Placebo Matching Escitalopram
  Arms: Placebo
Drug: Escitalopram — Active Escitalopram
  Arms: Escitalopram

SUMMARY:
The purpose is to determine if: 1) Escitalopram treatment will be associated with less oral corticosteroid use than placebo in outpatients with severe asthma and moderate or severe major depressive disorder (MDD). 2) Escitalopram treatment will be associated with greater improvement in asthma symptoms than placebo in outpatients with severe asthma and moderate or severe MDD. 3) Escitalopram treatment will be associated with greater depressive symptom remission rates than placebo in outpatients with severe asthma and moderate or severe MDD.

DETAILED DESCRIPTION:
Primary Aim

1) Determine if escitalopram treatment is associated with less oral corticosteroid use for asthma symptom control than placebo in asthma outpatients with moderate or MDD.

Secondary Aims

1. Determine if escitalopram treatment is associated with greater improvement in asthma symptoms than placebo in outpatients with severe asthma and moderate or severe MDD.
2. Determine if escitalopram treatment is associated with greater depressive symptom remission rates than placebo in outpatients with severe asthma and moderate or severe MDD.

Background/Significance

Asthma is a common, chronic general medical condition characterized by inflammation and variable, but usually reversible, airflow obstruction. Approximately 7.2% of people in the United States have a history of asthma. Asthma is common with an increasing prevalence and mortality especially in low-income and minority populations.

The course of asthma appears to be influenced by mood and emotions. It has been reported that there is a high prevalence of depression or depressive symptoms in both children and adults with asthma.

Depression is associated with increased use of asthma-related urgent care services, as well as a variety of unfavorable asthma outcomes. In addition to the possible associations between depression and asthma medication nonadherence and even death, depression appears to be associated with increased use of emergency rooms, hospitals, and unscheduled appointments for asthma.

Despite data on the frequency of depression in asthma and its adverse consequences, it is generally not recognized or treated.

Our proposed study is different. We observed a modest difference between antidepressant and placebo in a prior trial. However, in a subgroup with more severe asthma (based on frequent corticosteroid use) and more severe depression (based on higher depressive symptoms scores) we saw a much larger effect size. The proposed study will target this subgroup. The sample size is based on the effect size we observed in this subgroup in our previous pilot study.

A placebo controlled trial is needed because 1) the primary outcome in our previous trial was not significant. Therefore, it is not clear that antidepressant treatment is effective in depressed asthma patients. 2) We identified a subgroup with greater depressive symptom and asthma severity that based on a post-hoc analysis appeared to show a favorable response to the antidepressant. Thus, we want to confirm these post-hoc findings with a targeted prospective study. In the clinical population we will study, very few patients have ever received assessment or treatment for depression. Therefore, we would not be withholding clearly effective treatment that they would otherwise receive.

Standard of care for severe asthma is aggressive asthma treatment. Our study does not require any changes in the patient's asthma treatment. No guidelines are currently available on the treatment of depression in asthma patients. Standard care for depression would be antidepressants.

ELIGIBILITY:
Inclusion Criteria:

* Current HAM-D score of ≥ 20
* Patients with severe asthma (defined as asthma requiring three or more course of oral corticosteroids in the past year).
* No changes in asthma medications, oral corticosteroid use, or treatment for respiratory tract infections in the past week
* Needs to have taken ≥ 3 courses of oral corticosteroids, for asthma, in the past 12 months.
* Both male and female
* English- or Spanish-speaking

Exclusion Criteria:

* Current substance or alcohol abuse/dependence
* MDD with psychotic features (delusions, hallucinations, disorganized thought processes)
* Bipolar disorder
* Schizophrenia or schizoaffective disorder
* Substance-induced mood disorder and mood disorder secondary to a general medical condition
* Mental retardation or other severe cognitive impairment
* Prison or jail inmates
* Pregnant or nursing women or women of childbearing age who will not use The University of Texas Southwestern Medical Center - Institutional Review Board (UTSW IRB) approved methods of birth control or abstinence during the study
* Treatment-resistant depressed persons defined as having failed two adequate trials of antidepressants
* Current antipsychotic or antidepressant therapy or psychotherapy
* Initiation of other psychotropic medications or psychotherapy within past 2 weeks (e.g., anxiolytics, hypnotics)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Sherwood Brown, Ph.D, M.D., Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- The UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

REFERENCES:
- [Derived] Agarwal CD, Palka JM, Gajewski AJ, Khan DA, Brown ES. The efficacy of citalopram or escitalopram in patients with asthma and major depressive disorder. Ann Allergy Asthma Immunol. 2024 Mar;132(3):374-382. doi: 10.1016/j.anai.2023.11.004. Epub 2023 Nov 11. PMID 37952772

RESULTS

PARTICIPANT FLOW:
Groups:
- Matching Placebo: Placebo Matching Escitalopram taken orally daily (for a 12-week duration).
Period: Overall Study
Arm/Group | Escitalopram | Matching Placebo
Started | 13 | 13
Completed | 13 | 12
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: One participant had no post-baseline data, leaving 25 evaluable participants in the intent-to-treat sample that was used in the analysis.
Groups:
- Escitalopram: Active Escitalopram (A SSRI) taken orally in 10mg or 20mg doses daily.
- Placebo: Placebo Matching Escitalopram taken orally daily.
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Placebo | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (9.8) | 48.6 (12.7) | 45.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: HAM-D (Hamilton Rating Scale for Depression)
Description: The HAM-D is a 17 item questionnaire (a clinician-administered depression scale) designed to evaluate severity of depressive symptoms. Scores can range from 0 to 52. The higher the score, the worse the depressive symptoms (worse outcome).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale | 24.8 (4.4) | 28.3 (5.1)

2. Primary Outcome: ACQ (Asthma Control Questionnaire)
Description: The ACQ is a questionnaire used to assess symptoms pertinent to asthma management. Scores range from 0 to 42. The higher the score, the worse the asthma symptoms (worse outcome). The total ACQ score is obtained by dividing the raw score by the total number of items (in this case 7 items).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale | 1.9 (1.1) | 2.9 (0.9)

3. Primary Outcome: IDS-SR (Inventory of Depressive Symptomatology - Self-Report)
Description: The IDS-SR is a 30 item (self-report questionnaire) designed to assess symptoms of depression. Scores range from 0 to 90. The higher the score, the worse the depressive symptoms (worse outcome).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale | 35.2 (15.0) | 42.9 (12.3)

4. Primary Outcome: HAM-D (Hamilton Rating Scale for Depression)
Description: as for outcome 1
Time Frame: Up to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Matching Placebo: Placebo Matching Escitalopram taken orally daily.
Arm/Group | Escitalopram | Matching Placebo
Number analyzed (Participants) | 13 | 12
units on a scale | 16.7 (11.4) | 17.7 (7.6)

5. Primary Outcome: ACQ (Asthma Control Questionnaire)
Description: The ACQ is a questionnaire used to assess symptoms pertinent to asthma management.Scores range from 0 to 42. The higher the score, the worse the asthma symptoms (worse outcome). The total ACQ score is obtained by dividing the raw score by the total number of items (in this case 7 items).
Time Frame: Up to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram | Matching Placebo
Number analyzed (Participants) | 13 | 12
units on a scale | 1.9 (1.4) | 2.4 (1.2)

6. Primary Outcome: IDS-SR (Inventory of Depressive Symptomatology - Self-Report)
Description: as for outcome 3
Time Frame: Up to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram | Matching Placebo
Number analyzed (Participants) | 13 | 12
units on a scale | 26.3 (17.4) | 24.6 (14.9)

ADVERSE EVENTS:
Arm/Group | Escitalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 2/13 | 1/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (N=13) | Placebo (N=12)
Severe asthma attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Participant experienced a severe asthma attack, lost consciousness and was intubated at the intensive care unit. This event was serious, expected due to the patient's history, and not study-related. The patient was discontinued from the study.
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — This participant reported hospitalization for asthma exacerbation. This event was classified as serious, expected due to the patient's history, not study-related. The patient completed the study.
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — This participant was hospitalized for a worsening of asthma symptoms due to a viral respiratory infection that was successfully treated. This event was serious, unexpected, and not study-related. The patient was continued in the study.

LIMITATIONS AND CAVEATS:
A limitation of this proof-of-concept study was the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No